CLINICAL TRIAL: NCT03217006
Title: Randomized Comparison of the Clinical Outcome of Single Versus Multiple Arterial Grafts: the ROMA Trial
Brief Title: Randomization of Single vs Multiple Arterial Grafts
Acronym: ROMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1703018094; 1R01HL152021-01 (NIH)
Record Dates: First submitted 2017-07-06; First posted 2017-07-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease; Heart Diseases
Keywords: coronary artery bypass surgery; multiple arterial graft; radial artery graft
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Patients undergoing coronary artery bypass surgery will be in one of two groups. One group will receive a single arterial graft and the second group will receive two or more arterial grafts.
Who Masked: Outcomes Assessor
Masking Description: The endpoint assessors will be blinded to treatment allocation (PROBE).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Arterial Group (Experimental): Patients in this group will receive a single arterial graft which will be the left internal thoracic artery. Additional grafts used in this group will all be venous grafts.
  Interventions: Procedure: Single arterial graft
- Multiple Arterial Group (Experimental): Patients in the group will receive multiple arterial grafts. All patients will receive at least two arterial grafts, the left internal thoracic artery with the addition of either the right internal thoracic artery or the radial artery as the second conduit. Some patients may receive additional arterial grafts consisting of the radial artery, the right internal thoracic artery, or the right gastroepiploic artery.
  Interventions: Procedure: Multiple arterial grafting

INTERVENTIONS:
Procedure: Single arterial graft — This interventions consists of patients receiving the left internal thoracic artery to the left anterior descending coronary artery of the heart. In addition to the left internal thoracic artery patients will receive venous grafts for all additional grafting.
  Arms: Single Arterial Group
Procedure: Multiple arterial grafting — This intervention consists of the patient receiving the left internal thoracic artery to the left anterior descending coronary artery of the heart. The second arterial graft (right internal thoracic artery or radial artery) will be directed to the major branch of the circumflex. Additional grafts will include saphenous veins or arterial conduits.
  Arms: Multiple Arterial Group

SUMMARY:
The primary hypothesis of ROMA is that in patients undergoing primary isolated non-emergent coronary artery bypass surgery (CABG), the use of two or more arterial grafts compared to a single arterial graft is associated with a reduction in the composite outcome of death from any cause, any stroke, post discharge myocardial infarction and/or repeat revascularization. The secondary hypothesis is that in patients undergoing primary isolated non-emergent CABG, the use of two or more arterial grafts compared to a single arterial graft is associated with improved survival.

Prospective event-driven unblinded randomized multicenter trial of at least 4,300 subjects enrolled in at least 25 international centers. Patients will be randomized to a single arterial graft (SAG) or multiple arterial grafts (MAG). Patients will be randomized in a 1:1 fashion between the two groups. Permuted block randomization with random blocks stratified by the center and the type of second arterial graft will be used to provide treatment distribution in equal proportion.

DETAILED DESCRIPTION:
In the 1980's, it was recognized that long-term survival was enhanced in patients undergoing coronary surgery when the left anterior descending (LAD) was grafted with a left internal thoracic artery (ITA) rather than a saphenous vein (1). This difference was predicated, at least in part, due to greater and more durable patency of the left ITA compared to an increased early occlusion rate and later progressive atherosclerosis of saphenous vein grafts (SVG) (2).

For more than 20 years it has generally been accepted that patients who receive multiple arterial grafts (AGs) at the time of coronary artery bypass surgery (CABG) have increased postoperative survival compared to those who receive only one AG, especially over the long term (3-5). The current United States and European Guidelines encourage the use of AGs in patients with a long life expectancy (6, 7). Last year, a position paper from the Society of Thoracic Surgeons strongly recommended a wider use of AGs (8).

The putative mechanism underlying the AG hypothesis is greater patency. In line with the original findings of improved LAD graft patency with ITA vs. SVG, data from randomized control trials (RCTs) as well as observational studies and a network meta-analysis (9) have demonstrated that the patency of the RA, as well as the right ITA, exceed that of a SVG, providing mechanistic basis to support the AG hypothesis.

ROMA is a two arm event driven randomized multi-centre trial aimed at evaluating the impact of the use of one ITA vs two or more AGs for CABG on a composite of death from any cause, any stroke, post discharge myocardial infarction and/or repeat revascularization. The trial is powered to detect a 20% relative reduction in the primary outcome with 90% power at 5% alpha.

The primary aim is to conduct a multicenter international randomized control trial to test the hypothesis that the use of a two or more AGs compared to a single arterial graft is associated with a reduction in the composite outcome of death from any cause, any stroke, post discharge myocardial infarction and/or repeat revascularization.

The secondary aim is to conduct a multicenter international randomized control trial to test the hypothesis that the use of two or more AGs compared to a single arterial graft is associated with improved survival.

ELIGIBILITY:
Inclusion Criteria:

* Primary isolated CABG patients with disease of the left main coronary artery and/or of the left anterior descending and the circumflex coronary system with or without disease of the right coronary artery.

Exclusion Criteria:

* Age > 70 years
* Single graft
* Emergency operation
* Evolving myocardial infarction within 48 hours of surgery
* Left ventricular ejection fraction of < 35%
* Any concomitant cardiac or non-cardiac procedure
* Previous cardiac surgery
* Preoperative severe end-organ dysfunction (dialysis, liver failure, respiratory failure), cancer or any co-morbidity that reduce life expectancy to less than 5 years.
* Inability to use the saphenous vein or to use both radial and right internal thoracic arteries
* Anticipated need for coronary thrombo-endarterectomy
* Planned hybrid revascularization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4300 (Estimated)
Dates: Start 2018-01-07 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome | > 72 hours after surgery and/or repeat revascularization
  A composite of death from any cause, any stroke, post discharge myocardial infarction and/or repeat revascularization.

SECONDARY OUTCOMES:
30-day mortality | 30 days post-operatively
  Death from any cause at 30-days
Major postoperative complications | In-hospital stay, up to 30 days post-operatively
  Revision for bleeding, perioperative myocardial infarction, any stroke, need for dialysis, need for tracheostomy, and surgical site infection.
Sternal wound complication | 6 months post-operatively
  Wound drainage, skin separation, unstable sternum, and sternal dehiscence, infection
Composite Outcome of Death from any cause | Analysis will be performed after 631 events. The investigators assume this will occur at a mean follow-up of 5 years.
  A composite of death from any cause, post discharge myocardial infarction,stroke, and/or repeat revascularization
Stroke | Analysis will be performed after 631 events. The investigators assume this will occur at a mean follow-up of 5 years.
  Post discharge myocardial infarction and repeat revascularization considered as individual events
Cause-specific death (cardiac vs non-cardiac) | Analysis will be performed after 631 events. The investigators assume this will occur at a mean follow-up of 5 years
  Death as either cardiac or non-cardiac in etiology
Hospital readmissions | Analysis will be performed after 631 events. The investigators assume this will occur at a mean follow-up of 5 years
  Hospital readmissions with specific causes

CONTACTS AND LOCATIONS:
Overall Officials: Mario Gaudino, MD, Principal Investigator — Weill Medical College of Cornell University; Stephen Fremes, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (59):
- United States (11):
  - University of Colorado, Boulder, Colorado
  - Baystate Health, Springfield, Massachusetts
  - Nebraska Heart Hospital, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - Icahn School of Medicine, Mount Sinai, New York, New York
  - Weil Cornell Medical College Department of Cardiothoracic Surgery, New York, New York
  - Lenox Hill Hospital (Northwell), New York, New York
  - NewYork-Presbyterian Queens, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Allegheny General Hospital (Cardiovascular Institute), Pittsburgh, Pennsylvania
- Austria (3):
  - Innsbruck (Medical University) Austria, Innsbruck
  - Krankenhaus Nord Vienna North Hospital, Vienna
  - MU Vienna Austria, Vienna
- Federal University of Sao Paulo, São Paulo, Brazil
- Canada (9):
  - Hamilton General Hospital, Hamilton
  - London Health Sciences Ontario Canada, London
  - University Hospital of Montreal (CHUM), Montreal
  - University of Ottawa Heart Institute Canada, Ottawa
  - Royal Victoria Hospital (McGill), Québec
  - Universite Laval Quebec (CRIUCPQ) Canada, Québec
  - Sunnybrook Health Sciences Centre, Toronto
  - Toronto General Hospital, Toronto
  - St. Boniface General Hospital / WHRA, Winnipeg
- China (5):
  - Fuwai Hospital, Beijing
  - Jilin Heart Hospital, Changchun
  - Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - National Taiwan University Hospital, Taiwan
  - Teda Hospital (TICH), Tianjin
- University Hospital Dubrava, Zagreb, Croatia
- General University Hospital, Prague, Prague, Czechia
- Germany (11):
  - Duisburg Heart Center, Duisburg
  - Essen University, Duisburg
  - Düsseldorf University, Düsseldorf
  - University Hospital Erlangen, Erlangen
  - Giessen Hospital, Giessen
  - University Medical Center of Goettingen, Göttingen
  - Jena University Hospital, Jena
  - Heart Center (Herzzentrum), Leipzig
  - HDZ NRW Bad, Oeynhausen
  - Robert-Bosch-Hospital, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- Italy (6):
  - Anthea Hospital, Bari
  - Fondazione Poliambulanza, Brescia
  - Maria Cecilia Hospital GVM, Cotignola
  - Universita' Cattolica del Sacro Cuore, Roma
  - European Hospital, Rome
  - Ospedale Le Molinette, Torino
- Saitama Medical University, Saitama, Japan
- MUMC Maastricht (University Medical Centre), Maastricht, Netherlands
- Medical University of Silesia (Katowice), Katowice, Poland
- Portugal (3):
  - Hospitalar de Lisboa Central, Capuchos
  - University Hospital (Praceta Mota Pinto), Coimbra
  - Centro Hospitalar e Universitário São João, Porto
- Dedinje Cardiovascular Institute, Belgrade, Serbia
- National University of Singapore, Singapore, Singapore
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Sinchŏn-dong, South Korea
- Spain (2):
  - Hospital Univeritario Del Vinalopo, Alicante
  - Hospital Clinic de Barcelona (ICCV), Barcelona

REFERENCES:
- [Background] Loop FD, Lytle BW, Cosgrove DM, Stewart RW, Goormastic M, Williams GW, Golding LA, Gill CC, Taylor PC, Sheldon WC, et al. Influence of the internal-mammary-artery graft on 10-year survival and other cardiac events. N Engl J Med. 1986 Jan 2;314(1):1-6. doi: 10.1056/NEJM198601023140101. PMID 3484393
- [Background] Tatoulis J, Buxton BF, Fuller JA. Patencies of 2127 arterial to coronary conduits over 15 years. Ann Thorac Surg. 2004 Jan;77(1):93-101. doi: 10.1016/s0003-4975(03)01331-6. PMID 14726042
- [Background] Lytle BW, Blackstone EH, Loop FD, Houghtaling PL, Arnold JH, Akhrass R, McCarthy PM, Cosgrove DM. Two internal thoracic artery grafts are better than one. J Thorac Cardiovasc Surg. 1999 May;117(5):855-72. doi: 10.1016/S0022-5223(99)70365-X. PMID 10220677
- [Background] Taggart DP, D'Amico R, Altman DG. Effect of arterial revascularisation on survival: a systematic review of studies comparing bilateral and single internal mammary arteries. Lancet. 2001 Sep 15;358(9285):870-5. doi: 10.1016/S0140-6736(01)06069-X. PMID 11567701
- [Background] Yi G, Shine B, Rehman SM, Altman DG, Taggart DP. Effect of bilateral internal mammary artery grafts on long-term survival: a meta-analysis approach. Circulation. 2014 Aug 12;130(7):539-45. doi: 10.1161/CIRCULATIONAHA.113.004255. Epub 2014 Jun 10. PMID 24916209
- [Background] Hillis LD, Smith PK, Anderson JL, Bittl JA, Bridges CR, Byrne JG, Cigarroa JE, Disesa VJ, Hiratzka LF, Hutter AM Jr, Jessen ME, Keeley EC, Lahey SJ, Lange RA, London MJ, Mack MJ, Patel MR, Puskas JD, Sabik JF, Selnes O, Shahian DM, Trost JC, Winniford MD. 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 Dec 6;124(23):e652-735. doi: 10.1161/CIR.0b013e31823c074e. Epub 2011 Nov 7. No abstract available. PMID 22064599
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Aldea GS, Bakaeen FG, Pal J, Fremes S, Head SJ, Sabik J, Rosengart T, Kappetein AP, Thourani VH, Firestone S, Mitchell JD; Society of Thoracic Surgeons. The Society of Thoracic Surgeons Clinical Practice Guidelines on Arterial Conduits for Coronary Artery Bypass Grafting. Ann Thorac Surg. 2016 Feb;101(2):801-9. doi: 10.1016/j.athoracsur.2015.09.100. Epub 2015 Dec 8. PMID 26680310
- [Background] Benedetto U, Raja SG, Albanese A, Amrani M, Biondi-Zoccai G, Frati G. Searching for the second best graft for coronary artery bypass surgery: a network meta-analysis of randomized controlled trialsdagger. Eur J Cardiothorac Surg. 2015 Jan;47(1):59-65; discussion 65. doi: 10.1093/ejcts/ezu111. Epub 2014 Mar 30. PMID 24686003
- [Background] Nasso G, Coppola R, Bonifazi R, Piancone F, Bozzetti G, Speziale G. Arterial revascularization in primary coronary artery bypass grafting: Direct comparison of 4 strategies--results of the Stand-in-Y Mammary Study. J Thorac Cardiovasc Surg. 2009 May;137(5):1093-100. doi: 10.1016/j.jtcvs.2008.10.029. Epub 2009 Feb 7. PMID 19379973
- [Background] Taggart DP, Altman DG, Gray AM, Lees B, Gerry S, Benedetto U, Flather M; ART Investigators. Randomized Trial of Bilateral versus Single Internal-Thoracic-Artery Grafts. N Engl J Med. 2016 Dec 29;375(26):2540-9. doi: 10.1056/NEJMoa1610021. Epub 2016 Nov 14. PMID 27959712
- [Background] Zhang H, Wang ZW, Wu HB, Hu XP, Zhou Z, Xu P. Radial artery graft vs. saphenous vein graft for coronary artery bypass surgery : which conduit offers better efficacy? Herz. 2014 Jun;39(4):458-65. doi: 10.1007/s00059-013-3848-5. Epub 2013 Jun 21. PMID 23784362
- [Background] Harskamp RE, Alexander JH, Ferguson TB Jr, Hager R, Mack MJ, Englum B, Wojdyla D, Schulte PJ, Kouchoukos NT, de Winter RJ, Gibson CM, Peterson ED, Harrington RA, Smith PK, Lopes RD. Frequency and Predictors of Internal Mammary Artery Graft Failure and Subsequent Clinical Outcomes: Insights From the Project of Ex-vivo Vein Graft Engineering via Transfection (PREVENT) IV Trial. Circulation. 2016 Jan 12;133(2):131-8. doi: 10.1161/CIRCULATIONAHA.115.015549. Epub 2015 Dec 8. PMID 26647082
- [Background] Lopes RD, Mehta RH, Hafley GE, Williams JB, Mack MJ, Peterson ED, Allen KB, Harrington RA, Gibson CM, Califf RM, Kouchoukos NT, Ferguson TB Jr, Alexander JH; Project of Ex Vivo Vein Graft Engineering via Transfection IV (PREVENT IV) Investigators. Relationship between vein graft failure and subsequent clinical outcomes after coronary artery bypass surgery. Circulation. 2012 Feb 14;125(6):749-56. doi: 10.1161/CIRCULATIONAHA.111.040311. Epub 2012 Jan 11. PMID 22238227
- [Background] Shavadia J, Norris CM, Graham MM, Verma S, Ali I, Bainey KR. Symptomatic graft failure and impact on clinical outcome after coronary artery bypass grafting surgery: Results from the Alberta Provincial Project for Outcome Assessment in Coronary Heart Disease registry. Am Heart J. 2015 Jun;169(6):833-40. doi: 10.1016/j.ahj.2015.02.022. Epub 2015 Mar 13. PMID 26027621
- [Background] Gaudino M, Puskas JD, Di Franco A, Ohmes LB, Iannaccone M, Barbero U, Glineur D, Grau JB, Benedetto U, D'Ascenzo F, Gaita F, Girardi LN, Taggart DP. Three Arterial Grafts Improve Late Survival: A Meta-Analysis of Propensity-Matched Studies. Circulation. 2017 Mar 14;135(11):1036-1044. doi: 10.1161/CIRCULATIONAHA.116.025453. Epub 2017 Jan 24. PMID 28119382
- [Background] Yanagawa B, Verma S, Mazine A, Tam DY, Juni P, Puskas JD, Murugavel S, Friedrich JO. Impact of total arterial revascularization on long term survival: A systematic review and meta-analysis of 130,305 patients. Int J Cardiol. 2017 Apr 15;233:29-36. doi: 10.1016/j.ijcard.2017.02.010. Epub 2017 Feb 5. PMID 28185702
- [Background] Benedetto U, Gaudino M, Caputo M, Tranbaugh RF, Lau C, Di Franco A, Ng C, Girardi LN, Angelini GD. Right internal thoracic artery versus radial artery as the second best arterial conduit: Insights from a meta-analysis of propensity-matched data on long-term survival. J Thorac Cardiovasc Surg. 2016 Oct;152(4):1083-1091.e15. doi: 10.1016/j.jtcvs.2016.05.022. Epub 2016 May 28. PMID 27342731
- [Background] Hayward PA, Buxton BF. Mid-term results of the Radial Artery Patency and Clinical Outcomes randomized trial. Ann Cardiothorac Surg. 2013 Jul;2(4):458-66. doi: 10.3978/j.issn.2225-319X.2013.07.18. PMID 23977623
- [Background] Gaudino M, Cellini C, Pragliola C, Trani C, Burzotta F, Schiavoni G, Nasso G, Possati G. Arterial versus venous bypass grafts in patients with in-stent restenosis. Circulation. 2005 Aug 30;112(9 Suppl):I265-9. doi: 10.1161/CIRCULATIONAHA.104.512905. PMID 16159829
- [Background] Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, Mantel N, McPherson K, Peto J, Smith PG. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. I. Introduction and design. Br J Cancer. 1976 Dec;34(6):585-612. doi: 10.1038/bjc.1976.220. PMID 795448
- [Background] Serruys PW, Ong AT, van Herwerden LA, Sousa JE, Jatene A, Bonnier JJ, Schonberger JP, Buller N, Bonser R, Disco C, Backx B, Hugenholtz PG, Firth BG, Unger F. Five-year outcomes after coronary stenting versus bypass surgery for the treatment of multivessel disease: the final analysis of the Arterial Revascularization Therapies Study (ARTS) randomized trial. J Am Coll Cardiol. 2005 Aug 16;46(4):575-81. doi: 10.1016/j.jacc.2004.12.082. PMID 16098418
- [Derived] Masterson Creber R, Safford M, Ballman K, Myers A, Fremes S, Gaudino M. Randomized comparison of the clinical Outcome of single versus Multiple Arterial grafts: Quality of Life (ROMA:QOL) - Rationale and Study Protocol. Eur Heart J Qual Care Clin Outcomes. 2022 Aug 17;8(5):510-517. doi: 10.1093/ehjqcco/qcab022. PMID 33779716